CLINICAL TRIAL: NCT03450031
Title: Evaluation of Nasal Inflammatory Biomarkers During the Early and Late Phase Response to Nasal Volus Allergen Challenge in in Subjects With Seasonal Allergic Rhinitis (Out-of-season)
Brief Title: Evaluation of Nasal Inflammatory Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-13 XOBIO Pilot
Record Dates: First submitted 2018-01-30; First posted 2018-03-01 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC (no drug/no device) and NFP (Experimental): NAC with mixed grass pollen will be conducted. Nasal mucosal inflammatory mediators will be collected via nasal filter paper (NFP)
  Interventions: Other: NAC (no drug/no device)
- NAC (no drug/no device) and NFP AND NLF (Experimental): NAC with mixed grass pollen will be conducted. Nasal filter paper (NFP)sampling will be conducted from one nostril per time point. Subjects in Cohort B will also undergo nasal lavage (NLF) pre-NAC and at serial time points thereafter up to 8 hours
  Interventions: Other: NAC (no drug/no device)

INTERVENTIONS:
Other: NAC (no drug/no device) — Nasal allergen challenge (NAC) with mixed grass pollen: a bolus NAC with mixed grass pollen will be conducted

SUMMARY:
This research aims to establish a panel of inflammatory biomarkers of the early (Histamine, Tryptase, ProstaglandineD2) and late (Interleukin-4, Interleukin-5, Interleukin-6, Interleukin-13, Eotaxin, Tumor necrosis factor-a (TNF), (Macrophage Inflammatory Protein-1beta (MIP1ß)) phase response to nasal bolus allergen challenge (NAC) in subjects with out-of-season seasonal allergic rhinitis, suitable for future application in drug intervention studies of novel anti-allergy therapeutics.

DETAILED DESCRIPTION:
Biomarkers will be sampled by nasal filter paper (NFP) adsorption and lavage (NLF) prior to and following NAC. Samples from initial subjects (Cohort A; n~6) will be used primarily for validation of biomarker assays in nasal filter paper eluates. Validated biomarker assays will be applied to analyze biomarker changes in a further cohort of subjects (Cohort B; n~12) with the aim of fully defining the optimum panel and sampling time points for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent.
2. Male or female, age 18-65 years.

   Women will be considered for inclusion if they are:
   * Not pregnant, as confirmed by pregnancy test, and not nursing.
   * Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchal, or post-menopausal with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit).
   * Of childbearing potential and using a highly effective method of contraception during the entire study, as defined by at least one of the following

     * vasectomised partner
     * sexual abstinence (the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to Visit 2 procedures until at least 72 hours after NAC)
     * implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods (i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap)
3. History of seasonal allergic rhinitis to grass pollen with symptoms during the 2016 and 2017 allergen season requiring treatment with anti-histamines, nasal corticosteroids or leukotriene antagonists.
4. Absence of significant current symptoms of allergic rhinitis consistent with being out of season for their principal allergen (eg grass).
5. Skin prick test positive for mixed grass pollen allergen at Visit 1 or within one year prior to screening.

Exclusion criteria

1. Asthma requiring more than inhaled short-acting beta-2 agonists.
2. Spirometry showing FEV1 <80% predicted
3. Subjects who have smoked more than 5 cigarettes in the last 6 months or have a smoking history of ≥10 pack years.
4. Upper or lower respiratory tract infection in the prior 4 weeks.
5. Nasal or lung provocation procedure (eg, allergen challenge) conducted in the prior 4 weeks.
6. Significant nasal deformity, recent nasal surgery or obstructing nasal polyps.
7. History of anaphylaxis (any cause), or previous severe hypersensitivity reaction to any of the test agents for SPT or NAC.
8. Recent participation in a study of an investigational medicinal product (IMP) which could interfere with markers evaluated in this research
9. Use of any medications according to section 5.2 in the period indicated before Visit 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Interleukin-4 | Change from baseline at time points: 1 minutes (min), 4 min, 7 min, 10 min, 15 min, 30 min, 60 min, 120 min, 240 min, 360 min, 480 min
  Interlukin- 4 [pg/ml] using ELISA assays

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, Principal Investigator — Fraunhofer-Institute of Toxicology and Experimental Medicine
Locations (1):
- Fraunhofer ITEM im CRC, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No